CLINICAL TRIAL: NCT00021008
Title: A Phase II Open, Multicenter Trial to Assess the Activity and Tolerability of ZD0473 Given Intravenously as Second-line Therapy to Patients With Non-Small Lung Cancer Who Have Failed One Prior Platinum Based Chemotherapy Regimen
Brief Title: ZD0473 in Treating Patients With Progressive or Relapsed Non-Small Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068738; UCLA-000307201A; ZENECA-0473IL/0003; NCI-G01-1974
Record Dates: First submitted 2001-07-11; First posted 2004-04-13 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2001-09

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung | interventions — amminedichloro(2-methylpyridine)platinum(II)

INTERVENTIONS:
Drug: picoplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of ZD0473 in treating patients who have progressive or relapsed non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the anti-tumor effect of ZD0473 in patients with progressive or relapsed non-small cell lung cancer who have failed first-line platinum-based chemotherapy. II. Assess the safety and tolerability of this drug in these patients. III. Determine the pharmacokinetics of this drug in these patients. IV. Determine the efficacy of this drug, in terms of time to death, time to disease progression, disease control, and duration of response, in these patients. V. Assess the therapy outcome index, in terms of disease-related symptom relief, of these patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to time to relapse or progression after completion of first-line platinum-based chemotherapy (12 weeks or less vs more than 12 weeks). Patients receive ZD0473 IV over 1 hour on day 1. Treatment repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity. Quality of life is assessed at baseline, at the beginning of each course, and then every 6 weeks for 1 year after completion of study. Patients are followed at 30 days after study completion and every 6 weeks for 1 year.

PROJECTED ACCRUAL: A total of 32-73 patients (23-56 per stratum 1 and 9-17 per stratum 2) will be accrued for this study within approximately 9 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytologically confirmed non-small cell lung cancer Progressive or relapsed disease after first-line platinum-based chemotherapy Measurable disease No intracerebral metastases (unless asymptomatic, no corticosteroids required, and diagnostic imaging demonstrates no peritumoral edema or progression)

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: WHO 0-2 Life expectancy: More than 12 weeks Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hemoglobin at least 9 g/dL Hepatic: Bilirubin no greater than 1.25 times the upper limit of normal (ULN) ALT or AST less than 2.5 times ULN (5 times ULN if liver metastases present) No hepatic impairment No risk of hepatitis B transmission Renal: Creatinine clearance at least 60 mL/min Cardiovascular: No currently unstable or uncompensated cardiac conditions Pulmonary: No currently unstable or uncompensated respiratory conditions Other: No risk of HIV transmission No other malignancy within the past 5 years except adequately treated basal cell skin cancer or carcinoma in situ of the cervix No other severe or uncontrolled systemic disease No infectious condition No significant clinical disorder that would preclude study Body surface area at least 1.2 m2 Not pregnant or nursing Negative pregnancy test Fertile patients must use effective barrier contraception for 3 months before, during, and for 3 months after study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: See Disease Characteristics Radiotherapy: No prior extensive radiotherapy to 30% or more of bone marrow (e.g., whole of pelvis or half of spine) Surgery: Recovered from prior surgery Other: At least 2 weeks since prior systemic anticancer therapy and recovered

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Figlin, MD, FACP, Study Chair — Jonsson Comprehensive Cancer Center